CLINICAL TRIAL: NCT03073291
Title: Intervening to Prevent Youth Access to Marijuana Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Pacific Institute for Research and Evaluation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2R44DA038933-02 (NIH); 0309 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Cannabis
Keywords: cannabis; commerce
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of the psuedo-underage assessment of their retail recreational marijuana store. Pseudo-patron assessment teams will be unaware of the experimental condition to which each retail recreational marijuana store is assigned.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Responsible Marijuana Vendor Training (Experimental): The TrainToTend online responsible marijuana vendor training teaches responsible sales practices in five modules: Module 1, The Laws; Module 2, ID Checking; Module 3, Health Effects; Module 4, Customer Service, and Module 5, Rules of the Trade. The training content will be conveyed using online educational activities providing application and feedback such as in tabs with appropriate graphics and interactive simulations where users apply the skill and receive informative/corrective feedback.
  Interventions: Behavioral: Responsible Marijuana Vendor Training
- Usual and Customary Sales Practices Training (No Intervention): Usual and customary training in retail sales practices delivered to employees at retail recreational marijuana stores by store managers. Some retail stores in Colorado may receive responsible marijuana vendor training of some type from another state-approved training provider. Thus, we consider the outlets in the control group to have usual and customer sales training but not to be entirely untrained.

INTERVENTIONS:
Behavioral: Responsible Marijuana Vendor Training — Employees at retail recreational marijuana stores assigned to the the responsible marijuana vendor training will register them on TrainToTend online training program, create a user profile, and complete the training within four weeks from initial registration. Personnel who complete the training will receive a certificate of completion. New hires at the stores during the trial will be registered and complete the training within four weeks of commencing work. Separate versions of the training will be available reflecting differences in the laws/regulations on recreational marijuana sales in Colorado, Oregon, and Washington State and the content will be reviewed and approved by state regulators.
  Arms: Responsible Marijuana Vendor Training

SUMMARY:
The legalization of recreational marijuana use and sales in Alaska, Colorado, Oregon, and Washington State is a dramatic change in U.S. substance abuse policy that places a priority on developing regulatory and enforcement systems that prevent distribution of retail recreational marijuana to minors. Responsible marijuana vendor training, modeled after effective responsible alcoholic beverage training, has the potential to help the states prevent distribution to minors. This research will produce a responsible marijuana vendor training provided by a third party, not the cannabis industry, and test its effectiveness with retail recreational marijuana licensees and employees in Colorado, Oregon, and Washington State.

DETAILED DESCRIPTION:
The legalization of recreational marijuana in Alaska, Colorado, Oregon, and Washington State is the most dramatic change in U.S. substance abuse policy since the end of Prohibition. These states are implementing regulatory and enforcement systems for the retail sales of recreational marijuana to adults 21 years or older, akin to state controls on the sale of alcohol. In 2013, the U.S. Department of Justice (DOJ) issued directives that it would monitor whether these states implemented strong and effective regulatory and enforcement systems that among other DOJ priorities, prevented distribution of marijuana to youth. A retail sales intervention that has been effective at reducing illegal alcohol sales to minors (and intoxicated patrons) is alcoholic beverage server training (or responsible beverage service training). Recently, Colorado enacted a law for incentivized responsible marijuana vendor training, Oregon will require responsible marijuana vendor training, and Washington State may incentivize it. In this study, we propose to 1) produce the TrainToTend online responsible marijuana vendor training presenting retail marijuana sales laws, methods for checking IDs and preventing third party sales, the health effects of marijuana (e.g., fetal exposure; safe storage), customer service (e.g., driving under the influence; refusing sales to minors), and rules of the trade (e.g., inventory tracking and safety procedures) and 2) conduct a randomized trial on the TrainToTend training with a sample of retail recreational marijuana stores in Colorado, Oregon and Washington State (n=150) that are randomly assigned to have their employees complete the TrainToTend training (experimental group) or receive usual and customary sales training by store managers (no intervention control group). The effect of the TrainToTend training on responsible sales practices will be assessed by changes in recreational marijuana purchase attempts by pseudo-underage patrons (i.e., young-appearing customers without apparently valid IDs) at each store measured at 3-month follow-up and 9-month follow-up relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. being 21 or older,
2. owning a retail marijuana outlet or being employed as a manager or budtender at a retail marijuana outlet,
3. have a smart phone, tablet computer or personal computer with Internet access, and
4. consenting to participate

Exclusion Criteria:

1. a family or household member is already participating,
2. they are not proficient in English, or
3. they participated in the SBIR Phase I research

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Pseudo-underage Buyer Purchase Attempts | Baseline, 3-month follow-up, and 9-month follow-up
  Successful purchase attempts of a recreational marijuana product by underage-appearing pseudo-patron buyer will be assessed by pseudo-patron teams of a buyer and observer. The observer will enter the retail recreational marijuana store, showing a valid ID indicating they are 21 or older. The buyer will attempt to enter the store. If asked for an ID, the buyer will say they do not have a driver's license (acceptable form of ID) and offer instead a college ID (unacceptable form of ID). If permitted to enter store, buyer will ask to purchase pre-rolled joints. When the clerk asks the buyer to make payment, the buyer will say they do not have enough money and leave the store. The observer and buyer will record the outcome of the purchase attempt. No actual recreational marijuana product will be purchased.

SECONDARY OUTCOMES:
Change in State-required Store Signage | Baseline, 3-month follow-up, and 9-month follow-up
  Observers in the pseudo-patron teams will record the presence of signage in the stores required by state regulations.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Pacific Institute for Research and Evaluation, Oakland, California
  - Klein Buendel, Inc., Golden, Colorado

IPD SHARING:
Plan to Share IPD: No
At the conclusion of the project Klein Buendel Inc. will initiate a data sharing plan to make data from this project publicly available via archive files and publish reports describing study procedures in detail in peer-reviewed academic journals. Public data sets will be de-identified so that they are free of all identifiers that would permit linkages to individual research participants and of variables that could lead to deductive disclosure of the identity of individual participants. Individuals wishing to use this data will be required to fill out the KB Data Sharing Request Form, which asks for information on the type of data being requested, anticipated data use, research questions, study design, variables, analysis plan, and IRB approval.

REFERENCES:
- [Derived] Buller DB, Woodall WG, Saltz R, Grayson A, Buller MK, Cutter GR, Svendsen S, Liu X. Randomized Trial Testing an Online Responsible Vendor Training in Recreational Marijuana Stores in the United States. J Stud Alcohol Drugs. 2021 Mar;82(2):204-213. doi: 10.15288/jsad.2021.82.204. PMID 33823967
- [Derived] Buller DB, Woodall WG, Saltz R, Grayson A, Svendsen S, Cutter GR. Sales to apparently alcohol-intoxicated customers and online responsible vendor training in recreational cannabis stores in a randomized trial. Int J Drug Policy. 2020 Sep;83:102860. doi: 10.1016/j.drugpo.2020.102860. Epub 2020 Jul 21. PMID 32707476